CLINICAL TRIAL: NCT00753194
Title: False-Positive Results in Newborn Hearing Screening: Possible Causes
Brief Title: False Positive Results in Newborn Hearing Screening
Acronym: NHS
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Maria Cristina Silva simonek, Universidade Federal de Sao Paulo
Other Study IDs: 2612; 26129
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Deafness
Keywords: hearing; newborn; otoacoustic emissions
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Newborns that show a "Pass" On the newborn hearing screening program before hospital discharge
- 2: Newborns that show a "fail" and will be retested in 15 days.

SUMMARY:
The purpose of this study is to investigate the rate of false-positive results in Newborn Universal Hearing Screening Programs and it´s possible causes.

DETAILED DESCRIPTION:
False-positive results in Newborn Hearing Screening(NHS) leads to unnecessary parents anxiety and increase the cost of the procedure before hospital discharge. Getting to know the possible causes will lead to solutions to decrease the number of normal hearing babies that fail NHS with Otoacoustic Emissions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns

Exclusion Criteria:

* Risk factors for hearing loss

Ages: 6 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns
Sampling Method: Non-Probability Sample
Enrollment: 1110 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Otoacoustic Emissions | At birth

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Frasson, Doctor, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital Panamericano, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Grill E, Uus K, Hessel F, Davies L, Taylor RS, Wasem J, Bamford J. Neonatal hearing screening: modelling cost and effectiveness of hospital- and community-based screening. BMC Health Serv Res. 2006 Feb 23;6:14. doi: 10.1186/1472-6963-6-14. PMID 16504089
- See also: Non profitable organization that implemented Newborn Hearing Screening in Brazil — http://www.gatanu.org